CLINICAL TRIAL: NCT06134557
Title: Analysis of the Therapeutic Effect of Blood Flow Reconstruction in the Treatment of Intracranial Dissection Aneurysm of Vertebral Artery
Brief Title: Therapeutic Effect of Blood Flow Reconstruction in IVADA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202306-092
Record Dates: First submitted 2023-11-05; First posted 2023-11-18 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-11

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- flow diverter stents: single flow diverter(FD) stents or flow diverter assisted coil
  Interventions: Procedure: conventional stents
- conventional stents: stent-alone or overlapping stent treatment ,stent-assisted coiling techniques
  Interventions: Procedure: conventional stents

INTERVENTIONS:
Procedure: conventional stents — performed the study to compare the safety and efficacy between flow diverters and conventional stents in IVADA patients undergoing endovascular therapy. Stent-assisted coiling is the preferred option for most surgeons. In addition,It is believed that dense packing is not necessary as long as the aneurysm neck is covered to isolate the dissection. How ever,whether it is really necessary to adjunct coil,and if it is necesary, what is the ideal packing density of coils, there is no clear conclusion at present.This study aimed to compare the safety and efficacy between flow diverter and conventional stents in patients with IVADA, determine the ideal packing density of coils after FD stent placement,and to observe the hemodynamic changes before and after the treatment of FD stent.

SUMMARY:
IVADA (Intracranial vertebral artery dissecting aneurysms）is one of the causes of subarachnoid hemorrhage or posterior circulation ischemia with high mortality and disability. Current endovascular therapies for IVADA mainly include parent artery occlusion and endovascular blood reconstructive techniques. The method of parent artery occlusion requires the sacrifice of one vertebral artery. For the IVADA patients whose dissection involves PICA（posterior inferior cerebellar artery）or anterior spinal artery, severe ischemia even infarction of brain stem or cerebellar may be caused after parent artery occlusion , they are usually irreversible damage, so that method are rarely used now.Endovascular flood reconstructive techniques has become the mainstream, including stent-alone or overlapping stent treatment ,stent-assisted coiling techniques, single flow diverter(FD) stents or flow diverter assisted coil, etc.With the improvements in stents, flow diverter stent is efficient, while they are associated with the risk of ischemia, especially when vital arterial branches are covered. It has been reported that FD techniques have certain advantages over traditional stents in the treatment of anterior circulating intracranial aneurysms. In the treatment of posterior circulating aneurysms, perioperative ischemic complications increase due to their influence on the blood flow of perforator arteries, but there are few long-term observations at present. Currently, studies directly contrasting flow diverter and conventional stents in patients with IVADA are rare. Therefore, we performed the study to compare the safety and efficacy between flow diverters and conventional stents in IVADA patients undergoing endovascular therapy. Stent-assisted coiling is the preferred option for most surgeons. In addition,It is believed that dense packing is not necessary as long as the aneurysm neck is covered to isolate the dissection. How ever,whether it is really necessary to adjunct coil,and if it is necessary, what is the ideal packing density of coils, there is no clear conclusion at present.This study aimed to compare the safety and efficacy between flow diverter and conventional stents in patients with IVADA, determine the ideal packing density of coils after FD stent placement,and to observe the hemodynamic changes before and after the treatment of FD stent.

DETAILED DESCRIPTION:
This is a single-center, retrospective, and observational study.This retrospective study was approved by the Medical Ethics Committee of Qilu Hospital of Shandong University.Patients diagnosed with IVADA who underwent endovascular blood reconstructive treatment in the institution from December 2011 to December 2022 were eligible.Patient age, sex,index, clinical presentation, smoking, drinking, hypertension, diabetes mellitus, hyperlipidemia, modified Rankin Scale (mRS) score, aneurysm size, and arterial branch anatomy were recorded. Treatment details, complications, and angiographic and clinical outcomes were also recorded.

The optimal treatment strategy was evaluated based on the patients' neurological condition and comorbidities, the angioarchitectural features of the aneurysm, and the decision of the patient and their first degree relatives. The conventional stents included Neuroform (Stryker Neurovascular, USA), Enterprise (Cordis Neurovascular, USA), and Solitaire (ev3, USA) stents, and a low-profile visualized intraluminal support (LVIS) device (MicroVention Terumo, USA) was used. The flow diverters included Tubridge (MicroPort NeuroTech, China) and Pipeline (Medtronic, USA) devices. All EVT procedures were performed via a femoral artery approach under general anesthesia. An intravenous bolus of heparin (5000 IU) was administered before the procedure. Heparin was discontinued at the end of the procedure. A standard 6F or 8F guide catheter was advanced into the subclavian artery, proximal to the vertebral artery. An intermediate catheter (Navien, Medtronic) was then inserted into the V2 segment of the vertebral artery. A stent microcatheter was used to access the true lumen of the aneurysm in the posterior cerebral artery through the guidewire. For cases with additional coil insertion, a coil microcatheter was placed in the aneurysm sac. The stent was partially deployed to cover the aneurysm neck and temporarily jail the microcatheter, after which the aneurysm was loosely or densely packed with detachable coils before the stent was completely deployed. For long segmental lesions in which the aneurysm neck could not be covered completely with a single stent, an additional stent was extended into the bridged segment. If a single stent was not sufficient to alter the intra-aneurysmal hemodynamics, overlapping stents were used to reconstruct the lesion.

The anti-platelet drugs (aspirin 100 mg/day and clopidogrel 75 mg/day) were administered for at least 3 days prior to the procedure for patients with unruptured aneurysms. All patients with ruptured aneurysm were given aspirin and clopidogrel 300mg by oral or nasal feeding before general anesthesia was administered.The anti-platelet drugs (aspirin 100 mg/day and clopidogrel 75 mg/day) were administered for 3 months post-operatively, followed by aspirin alone for 3 months. Patients who had insufficient responses to aspirin or clopidogrel received a substitute antiplatelet agent (ticagrelor).The diameter and length of the stent were chosen according to the dimensions of the affected parent vessel.

The main complications during hospitalization were hemorrhage, infarction, or hydrocephalus requiring shunting. Procedural complications included those that occurred intraoperatively or after EVT. Periprocedural complications included those that occurred during hospitalization. Clinical follow-up was performed via neurological examinations or telephone interviews. Clinical outcomes were assigned based on the modified Rankin scale (mRS) score at the last follow-up: 0-2, favorable outcome; 3-6, unfavorable outcome. Cerebral angiography was performed at 6 months after EVT to confirm aneurysm occlusion and the patency of the VA（vertebral artery）. Aneurysm occlusions on immediate and final follow-up cerebral angiography were categorized as complete occlusion (no filling of the contrast agent in the aneurysm sac) or incomplete occlusion (residual filling of the contrast agent in the aneurysm neck or sac).

Imaging follow-up was performed using DSA（digital subtraction angiography）、CTA（Computer Tomographic Angiography）、MRA（Magnetic Resonance Angiography） approximately 6 months after stenting. The occlusion rate was evaluated using the O'KellyMarotta (OKM) grading scale . Recurrence was defined as an aneurysm that showed an increased percentage of contrast filling within the aneurysmal sac on follow-up angiography. All imaging studies were evaluated independently by two neurointerventionalists with more than 5 years of experience. Any disagreements were resolved by third neurointerventionalists with 10 years of experience. Clinical outcomes were evaluated by determining the mRS score at follow-up visits or via telephone interviews.

Using The R Programming Language software,Propensity Score Matching 1：2 (caliper value 0.05), to make it has no statistical differences between the two groups in baseline information. The matched case data will be statistically analyzed by IBM SPSS Statistics27.0(IBM Corp, New York, USA)。 The one-sample Kolmogorov-Smirnov test was used to test the normality of the data distribution for continuous variables. Continuous variables that conforming to a normal distribution are presented as mean and SD, and do not conform to the normal distribution are expressed by the median (25%,75%).Categorical variables are presented as numbers (frequency). Continuous variables were compared using the Student's t-test or Mann-Whitney U test, as appropriate. Categorical variables were compared using the chi-square test or Fisher's exact test, as appropriate. Variables identified as potential predictors in univariate analysis (p<0.1) were included in binary logistic regression analysis (forward) to determine their status as independent predictors. A p value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with asymptomatic or SAH symptoms of intracranial hypertension
2. After a preliminary diagnosis of cerebrovascular CTA or MRA, DSA angiography confirmed IVADA
3. IVADA involves intracranial segment of vertebral artery (V4 )

Exclusion Criteria:

* : Patients with SAH caused by trauma or other cerebrovascular diseases

  2: IVADA involves the extracranial vertebral artery

  3: Vertebrobasilar artery tortuosity and dilatation

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IVADA who underwent endovascular blood reconstructive tratement in our institution
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
complete aneurysm occlusion | 6 months postoperatively
  whether obtain complete aneurysm occlusion
Complications | during hospitalization（up to day 3） and post-discharge（12months post-discharge）
  Ischemic or hemorrhagic complications

CONTACTS AND LOCATIONS:
Overall Officials: Yunyan Wang, Study Chair — Medical Ethics Committee of Qilu Hospital of Shandong University; Weiying Zhong, Study Director — Medical Ethics Committee of Qilu Hospital of Shandong University; Maogui li, Principal Investigator — Medical Ethics Committee of Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Suzuki H, Kitagawa T, Gotoh M, Mitsueda-Ono T, Matsui M. Cervical Cord Infarction Caused by Dissection of the Intracranial Segment of the Vertebral Artery. Intern Med. 2018 Nov 15;57(22):3321-3324. doi: 10.2169/internalmedicine.0608-17. Epub 2018 Jul 6. PMID 29984769
- [Result] Debette S, Compter A, Labeyrie MA, Uyttenboogaart M, Metso TM, Majersik JJ, Goeggel-Simonetti B, Engelter ST, Pezzini A, Bijlenga P, Southerland AM, Naggara O, Bejot Y, Cole JW, Ducros A, Giacalone G, Schilling S, Reiner P, Sarikaya H, Welleweerd JC, Kappelle LJ, de Borst GJ, Bonati LH, Jung S, Thijs V, Martin JJ, Brandt T, Grond-Ginsbach C, Kloss M, Mizutani T, Minematsu K, Meschia JF, Pereira VM, Bersano A, Touze E, Lyrer PA, Leys D, Chabriat H, Markus HS, Worrall BB, Chabrier S, Baumgartner R, Stapf C, Tatlisumak T, Arnold M, Bousser MG. Epidemiology, pathophysiology, diagnosis, and management of intracranial artery dissection. Lancet Neurol. 2015 Jun;14(6):640-54. doi: 10.1016/S1474-4422(15)00009-5. PMID 25987283
- [Result] Mizutani T, Aruga T, Kirino T, Miki Y, Saito I, Tsuchida T. Recurrent subarachnoid hemorrhage from untreated ruptured vertebrobasilar dissecting aneurysms. Neurosurgery. 1995 May;36(5):905-11; discussion 912-3. doi: 10.1227/00006123-199505000-00003. PMID 7791980
- [Result] Gottesman RF, Sharma P, Robinson KA, Arnan M, Tsui M, Saber-Tehrani A, Newman-Toker DE. Imaging characteristics of symptomatic vertebral artery dissection: a systematic review. Neurologist. 2012 Sep;18(5):255-60. doi: 10.1097/NRL.0b013e3182675511. PMID 22931729
- [Result] Han M, Rim NJ, Lee JS, Kim SY, Choi JW. Feasibility of high-resolution MR imaging for the diagnosis of intracranial vertebrobasilar artery dissection. Eur Radiol. 2014 Dec;24(12):3017-24. doi: 10.1007/s00330-014-3296-5. Epub 2014 Jul 14. PMID 25017728
- [Result] Zang YZ, Wang ZG, Wang CW, Zhang Y, Ding X, Wang XF. [Clinical analysis of endovascular strategies in the treatment of vertebrobasilar dissecting aneurysms]. Zhonghua Yi Xue Za Zhi. 2016 Nov 8;96(41):3329-3332. doi: 10.3760/cma.j.issn.0376-2491.2016.41.011. Chinese. PMID 27852380
- [Result] Kim BM, Shin YS, Baik MW, Lee DH, Jeon P, Baik SK, Lee TH, Kang DH, Suh SI, Byun JS, Jung JY, Kwon K, Kim DJ, Park KY, Kim BS, Park JC, Kim SR, Kim YW, Kim H, Jo K, Yoon CH, Kim YS. Pipeline Embolization Device for Large/Giant or Fusiform Aneurysms: An Initial Multi-Center Experience in Korea. Neurointervention. 2016 Mar;11(1):10-7. doi: 10.5469/neuroint.2016.11.1.10. Epub 2016 Mar 3. PMID 26958407
- [Result] Acke F, Acou M, Hemelsoet D. Basilar artery dissection. Acta Neurol Belg. 2011 Dec;111(4):376. No abstract available. PMID 22368989
- [Result] Conforto AB. Challenges in diagnosis and treatment of cervico-cephalic arterial dissections. Arq Neuropsiquiatr. 2016 Apr;74(4):273-4. doi: 10.1590/0004-282X20160039. No abstract available. PMID 27096998
- [Result] Choi JW, Han DH, Kang KD, Jung HY, Renshaw PF. Aerobic exercise and attention deficit hyperactivity disorder: brain research. Med Sci Sports Exerc. 2015 Jan;47(1):33-9. doi: 10.1249/MSS.0000000000000373. PMID 24824770
- [Result] Wang Y, Cui L, Ji X, Dong Q, Zeng J, Wang Y, Zhou Y, Zhao X, Wang C, Liu L, Nguyen-Huynh MN, Claiborne Johnston S, Wong L, Li H; China National Stroke Registry Investigators. The China National Stroke Registry for patients with acute cerebrovascular events: design, rationale, and baseline patient characteristics. Int J Stroke. 2011 Aug;6(4):355-61. doi: 10.1111/j.1747-4949.2011.00584.x. Epub 2011 Feb 17. PMID 21609414
- [Result] Bejot Y, Daubail B, Debette S, Durier J, Giroud M. Incidence and outcome of cerebrovascular events related to cervical artery dissection: the Dijon Stroke Registry. Int J Stroke. 2014 Oct;9(7):879-82. doi: 10.1111/ijs.12154. Epub 2013 Oct 22. PMID 24148660
- [Result] Kapsalaki EZ, Rountas CD, Fountas KN. The Role of 3 Tesla MRA in the Detection of Intracranial Aneurysms. Int J Vasc Med. 2012;2012:792834. doi: 10.1155/2012/792834. Epub 2012 Jan 16. PMID 22292121
- [Result] Balik V, Yamada Y, Talari S, Kei Y, Sano H, Suyama D, Kawase T, Takagi K, Takizawa K, Kato Y. State-of-art in surgical treatment of dissecting posterior circulation intracranial aneurysms. Neurosurg Rev. 2018 Jan;41(1):31-45. doi: 10.1007/s10143-016-0749-0. Epub 2016 May 24. PMID 27215913
- [Result] Darsaut TE, Findlay JM, Magro E, Kotowski M, Roy D, Weill A, Bojanowski MW, Chaalala C, Iancu D, Lesiuk H, Sinclair J, Scholtes F, Martin D, Chow MM, O'Kelly CJ, Wong JH, Butcher K, Fox AJ, Arthur AS, Guilbert F, Tian L, Chagnon M, Nolet S, Gevry G, Raymond J. Surgical clipping or endovascular coiling for unruptured intracranial aneurysms: a pragmatic randomised trial. J Neurol Neurosurg Psychiatry. 2017 Aug;88(8):663-668. doi: 10.1136/jnnp-2016-315433. Epub 2017 Jun 20. PMID 28634280
- [Result] Shi L, Xu K, Sun X, Yu J. Therapeutic Progress in Treating Vertebral Dissecting Aneurysms Involving the Posterior Inferior Cerebellar Artery. Int J Med Sci. 2016 Jun 30;13(7):540-55. doi: 10.7150/ijms.15233. eCollection 2016. PMID 27429591
- [Result] Ortiz J, Ruland S. Cervicocerebral artery dissection. Curr Opin Cardiol. 2015 Nov;30(6):603-10. doi: 10.1097/HCO.0000000000000224. PMID 26447501
- [Result] Sonmez O, Brinjikji W, Murad MH, Lanzino G. Deconstructive and Reconstructive Techniques in Treatment of Vertebrobasilar Dissecting Aneurysms: A Systematic Review and Meta-Analysis. AJNR Am J Neuroradiol. 2015 Jul;36(7):1293-8. doi: 10.3174/ajnr.A4360. Epub 2015 May 7. PMID 25953763
- [Result] Ohta H, Natarajan SK, Hauck EF, Khalessi AA, Siddiqui AH, Hopkins LN, Levy EI. Endovascular stent therapy for extracranial and intracranial carotid artery dissection: single-center experience. J Neurosurg. 2011 Jul;115(1):91-100. doi: 10.3171/2011.1.JNS091806. Epub 2011 Mar 18. PMID 21417710
- [Result] Wang Y, Zhao C, Hao X, Wang C, Wang Z. Endovascular interventional therapy and classification of vertebral artery dissecting aneurysms. Exp Ther Med. 2014 Nov;8(5):1409-1415. doi: 10.3892/etm.2014.1961. Epub 2014 Sep 12. PMID 25289031
- [Result] Park W, Ahn JS, Park JC, Kwun BD, Kim CJ. Occipital artery-posterior inferior cerebellar artery bypass for the treatment of aneurysms arising from the vertebral artery and its branches. World Neurosurg. 2014 Nov;82(5):714-21. doi: 10.1016/j.wneu.2014.06.053. Epub 2014 Jul 3. PMID 24998497
- [Result] Lylyk P, Ceratto R, Hurvitz D, Basso A. Treatment of a vertebral dissecting aneurysm with stents and coils: technical case report. Neurosurgery. 1998 Aug;43(2):385-8. doi: 10.1097/00006123-199808000-00132. PMID 9696097
- [Result] Suzuki S, Kurata A, Iwamoto K, Sato K, Niki J, Miyazaki T, Yamada M, Oka H, Fujii K, Kan S. Endovascular surgery using stents for vertebral artery dissecting aneurysms and a review of the literature. Minim Invasive Neurosurg. 2008 Aug;51(4):193-8. doi: 10.1055/s-2008-1073172. PMID 18683108
- [Result] Li H, Gao BL, Li CH, Wang JW, Liu JF, Yang ST. Endovascular Retreatment of Cerebral Aneurysms Previously Treated with Endovascular Embolization. J Neurol Surg A Cent Eur Neurosurg. 2020 May;81(3):207-212. doi: 10.1055/s-0039-1685513. Epub 2019 Nov 19. PMID 31746449
- [Result] Chalouhi N, Tjoumakaris S, Gonzalez LF, Dumont AS, Starke RM, Hasan D, Wu C, Singhal S, Moukarzel LA, Rosenwasser R, Jabbour P. Coiling of large and giant aneurysms: complications and long-term results of 334 cases. AJNR Am J Neuroradiol. 2014 Mar;35(3):546-52. doi: 10.3174/ajnr.A3696. Epub 2013 Aug 14. PMID 23945229
- [Result] Endo H, Matsumoto Y, Kondo R, Sato K, Fujimura M, Inoue T, Shimizu H, Takahashi A, Tominaga T. Medullary infarction as a poor prognostic factor after internal coil trapping of a ruptured vertebral artery dissection. J Neurosurg. 2013 Jan;118(1):131-9. doi: 10.3171/2012.9.JNS12566. Epub 2012 Oct 5. PMID 23039149
- [Result] Khattak YJ, Sibaie AA, Anwar M, Sayani R. Stents and Stent Mimickers in Endovascular Management of Wide-neck Intracranial Aneurysms. Cureus. 2018 Oct 5;10(10):e3420. doi: 10.7759/cureus.3420. PMID 30542634
- [Result] Liu J, Li X, Sun S, Wang Y, Zang P. Clinical and Angiographic Outcomes of Endovascular Treatment for Ruptured Posterior Circulation Cerebral Aneurysms. Turk Neurosurg. 2016;26(4):513-7. doi: 10.5137/1019-5149.JTN.6570-12.1. PMID 27400096
- [Result] Iannaccone Farkasova S, Sopkova D, Svajdler M Jr, Farkas D, Mistrikova L, Mezencev R. Chronic dissecting aneurysm of ascending aorta with a large intramural thrombus and isolated aortic defects. Cesk Patol. 2019 Spring;55(2):115-119. PMID 31181944
- [Result] Jin SC, Kwon DH, Choi CG, Ahn JS, Kwun BD. Endovascular strategies for vertebrobasilar dissecting aneurysms. AJNR Am J Neuroradiol. 2009 Sep;30(8):1518-23. doi: 10.3174/ajnr.A1621. Epub 2009 May 27. PMID 19474118
- [Result] Marosfoi M, Langan ET, Strittmatter L, van der Marel K, Vedantham S, Arends J, Lylyk IR, Loganathan S, Hendricks GM, Szikora I, Puri AS, Wakhloo AK, Gounis MJ. In situ tissue engineering: endothelial growth patterns as a function of flow diverter design. J Neurointerv Surg. 2017 Oct;9(10):994-998. doi: 10.1136/neurintsurg-2016-012669. Epub 2016 Oct 5. PMID 27707872
- [Result] Brinjikji W, Murad MH, Lanzino G, Cloft HJ, Kallmes DF. Endovascular treatment of intracranial aneurysms with flow diverters: a meta-analysis. Stroke. 2013 Feb;44(2):442-7. doi: 10.1161/STROKEAHA.112.678151. Epub 2013 Jan 15. PMID 23321438
- [Result] Kan P, Sweid A, Srivatsan A, Jabbour P. Expanding Indications for Flow Diverters: Ruptured Aneurysms, Blister Aneurysms, and Dissecting Aneurysms. Neurosurgery. 2020 Jan 1;86(Suppl 1):S96-S103. doi: 10.1093/neuros/nyz304. PMID 31838529
- [Result] Deng Q, Feng W, Hai H, Liu J. Evaluation of the safety and efficacy of a Pipeline Flex embolization device for treatment of large, wide-necked intracranial aneurysms. J Interv Med. 2019 Apr 30;1(4):229-233. doi: 10.19779/j.cnki.2096-3602.2018.04.06. eCollection 2018 Nov. PMID 34805855
- [Result] Adeeb N, Griessenauer CJ, Dmytriw AA, Shallwani H, Gupta R, Foreman PM, Shakir H, Moore J, Limbucci N, Mangiafico S, Kumar A, Michelozzi C, Zhang Y, Pereira VM, Matouk CC, Harrigan MR, Siddiqui AH, Levy EI, Renieri L, Marotta TR, Cognard C, Ogilvy CS, Thomas AJ. Risk of Branch Occlusion and Ischemic Complications with the Pipeline Embolization Device in the Treatment of Posterior Circulation Aneurysms. AJNR Am J Neuroradiol. 2018 Jul;39(7):1303-1309. doi: 10.3174/ajnr.A5696. Epub 2018 Jun 7. PMID 29880475
- [Result] Wang K, Tian Z, Chen J, Liu J, Wang Y, Zhang H, Wang J, Zhang Y, Yang X. Risk Factors of Recurrence after Stent(s)-Assisted Coiling of Intracranial Vertebrobasilar Dissecting Aneurysms: A Multicenter Study. Front Neurol. 2017 Sep 14;8:482. doi: 10.3389/fneur.2017.00482. eCollection 2017. PMID 28959233
- [Result] Cagnazzo F, Perrini P, Dargazanli C, Lefevre PH, Gascou G, Morganti R, di Carlo D, Derraz I, Riquelme C, Bonafe A, Costalat V. Treatment of Unruptured Distal Anterior Circulation Aneurysms with Flow-Diverter Stents: A Meta-Analysis. AJNR Am J Neuroradiol. 2019 Apr;40(4):687-693. doi: 10.3174/ajnr.A6002. Epub 2019 Mar 14. PMID 30872418
- [Result] Bender MT, Colby GP, Jiang B, Lin LM, Campos JK, Xu R, Westbroek EM, Vo CD, Zarrin DA, Caplan JM, Huang J, Tamargo RJ, Coon AL. Flow Diversion of Posterior Circulation Cerebral Aneurysms: A Single-Institution Series of 59 Cases. Neurosurgery. 2019 Jan 1;84(1):206-216. doi: 10.1093/neuros/nyy076. PMID 29608702
- [Result] Griessenauer CJ, Ogilvy CS, Adeeb N, Dmytriw AA, Foreman PM, Shallwani H, Limbucci N, Mangiafico S, Kumar A, Michelozzi C, Krings T, Pereira VM, Matouk CC, Harrigan MR, Shakir HJ, Siddiqui AH, Levy EI, Renieri L, Marotta TR, Cognard C, Thomas AJ. Pipeline embolization of posterior circulation aneurysms: a multicenter study of 131 aneurysms. J Neurosurg. 2019 Mar 1;130(3):923-935. doi: 10.3171/2017.9.JNS171376. Epub 2018 May 4. PMID 29726768
- [Result] Albuquerque FC, Park MS, Abla AA, Crowley RW, Ducruet AF, McDougall CG. A reappraisal of the Pipeline embolization device for the treatment of posterior circulation aneurysms. J Neurointerv Surg. 2015 Sep;7(9):641-5. doi: 10.1136/neurintsurg-2014-011340. Epub 2014 Aug 4. PMID 25092926
- [Result] Lopes DK, Jang DK, Cekirge S, Fiorella D, Hanel RA, Kallmes DF, Levy EI, Lylyk P. Morbidity and Mortality in Patients With Posterior Circulation Aneurysms Treated With the Pipeline Embolization Device: A Subgroup Analysis of the International Retrospective Study of the Pipeline Embolization Device. Neurosurgery. 2018 Sep 1;83(3):488-500. doi: 10.1093/neuros/nyx467. PMID 28945879
- [Result] Kuhn AL, Kan P, Massari F, Lozano JD, Hou SY, Howk M, Gounis MJ, Wakhloo AK, Puri AS. Endovascular reconstruction of unruptured intradural vertebral artery dissecting aneurysms with the Pipeline embolization device. J Neurointerv Surg. 2016 Oct;8(10):1048-51. doi: 10.1136/neurintsurg-2015-012028. Epub 2015 Nov 6. PMID 26546600
- [Result] Fischer S, Perez MA, Kurre W, Albes G, Bazner H, Henkes H. Pipeline embolization device for the treatment of intra- and extracranial fusiform and dissecting aneurysms: initial experience and long-term follow-up. Neurosurgery. 2014 Oct;75(4):364-74; discussion 374. doi: 10.1227/NEU.0000000000000431. PMID 24871140
- [Result] Corley JA, Zomorodi A, Gonzalez LF. Treatment of Dissecting Distal Vertebral Artery (V4) Aneurysms With Flow Diverters. Oper Neurosurg. 2018 Jul 1;15(1):1-9. doi: 10.1093/ons/opx180. PMID 28962011
- [Result] Tan LA, Moftakhar R, Lopes DK. Treatment of a ruptured vertebrobasilar fusiform aneurysm using pipeline embolization device. J Cerebrovasc Endovasc Neurosurg. 2013 Mar;15(1):30-3. doi: 10.7461/jcen.2013.15.1.30. Epub 2013 Mar 31. PMID 23593603
- [Result] Narata AP, Yilmaz H, Schaller K, Lovblad KO, Pereira VM. Flow-diverting stent for ruptured intracranial dissecting aneurysm of vertebral artery. Neurosurgery. 2012 Apr;70(4):982-8; discussion 988-9. doi: 10.1227/NEU.0b013e318236715e. PMID 21937937
- [Result] Guerrero WR, Ortega-Gutierrez S, Hayakawa M, Derdeyn CP, Rossen JD, Hasan D, Samaniego EA. Endovascular Treatment of Ruptured Vertebrobasilar Dissecting Aneurysms Using Flow Diversion Embolization Devices: Single-Institution Experience. World Neurosurg. 2018 Jan;109:e164-e169. doi: 10.1016/j.wneu.2017.09.125. Epub 2017 Oct 5. PMID 28987840
- [Result] Maus V, Mpotsaris A, Dorn F, Mohlenbruch M, Borggrefe J, Stavrinou P, Abdullayev N, Barnikol UB, Liebig T, Kabbasch C. The Use of Flow Diverter in Ruptured, Dissecting Intracranial Aneurysms of the Posterior Circulation. World Neurosurg. 2018 Mar;111:e424-e433. doi: 10.1016/j.wneu.2017.12.095. Epub 2017 Dec 23. PMID 29277587
- [Result] Lin N, Brouillard AM, Krishna C, Mokin M, Natarajan SK, Sonig A, Snyder KV, Levy EI, Siddiqui AH. Use of coils in conjunction with the pipeline embolization device for treatment of intracranial aneurysms. Neurosurgery. 2015 Feb;76(2):142-9. doi: 10.1227/NEU.0000000000000579. PMID 25255261
- [Result] Chong W, Zhang Y, Qian Y, Lai L, Parker G, Mitchell K. Computational hemodynamics analysis of intracranial aneurysms treated with flow diverters: correlation with clinical outcomes. AJNR Am J Neuroradiol. 2014 Jan;35(1):136-42. doi: 10.3174/ajnr.A3790. Epub 2013 Nov 28. PMID 24287091
- [Derived] Zhang T, Zhong W, Zhou D, Xu Y, Li M, Zhuang J, Wang D, Su W, Wang Y. Treatment of unruptured intracranial vertebral artery dissection aneurysms with Flow Diverter compared with conventional stent-assisted coiling-a single-center study. Acta Neurochir (Wien). 2024 Dec 18;166(1):506. doi: 10.1007/s00701-024-06398-z. PMID 39690339